CLINICAL TRIAL: NCT05852795
Title: Evaluating the Behavioral Effect of a Virtual Reality-mediated Mindfulness-based Interventions on Parents of Children With Autism: a Randomized Controlled Trial (RCT) Study
Brief Title: Virtual Reality Experiences as Tools to Support Mental Health in Parents of Children With Autism
Acronym: Mind-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Antonio Cerasa, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CNR-IRIB-PRO-2023-001
Record Dates: First submitted 2023-04-24; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder; Parents
Keywords: Autism; Parents; Virtual Reality; Mental health; Mindfulness; Parental wellbeing
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): VR-based and audio-based mindfulness experience. Partecipants watch VR scenario and receive a guided mindfulness practice.
  Interventions: Other: Virtual Reality-mediated Mindfulness-Based Interventions
- Control Group (Other): VR-based mindfulness experience. Participants watch VR scenario without experiencing voice guided mindfulness practice.
  Interventions: Other: Virtual Reality-mediated Mindfulness-Based Interventions without audio guided experience

INTERVENTIONS:
Other: Virtual Reality-mediated Mindfulness-Based Interventions — The Experimental will undergo 8 weekly sessions of immersive experience lasting 30 minutes. Each session is divided as follows:
  * First phase: Detection of physiological parameters with Oculus equipment switched off (10 minutes).
  * Second phase: Detection of physiological parameters with Oculus instrumentation turned ON during mindfulness experience (10 minutes
  * Third phase: Detection of physiological parameters with Oculus equipment switched off (10 minutes).
  This intervention will produce a multisensory experience merging visual and digital auditory stimuli. The audio recording also included some ambient natural sound effects, to make the practice more immersive.
  Arms: Experimental group
Other: Virtual Reality-mediated Mindfulness-Based Interventions without audio guided experience — The Control will undergo 8 weekly sessions of immersive experience lasting 30 minutes. Each session is divided as follows:
  * First phase: Detection of physiological parameters with Oculus equipment switched off (10 minutes).
  * Second phase: Detection of physiological parameters with Oculus instrumentation turned ON during mindfulness experience (10 minutes
  * Third phase: Detection of physiological parameters with Oculus equipment switched off (10 minutes).
  This intervention will produce a monosensorial experience with video guided stimulation of naturalistic scenarios.
  Arms: Control Group

SUMMARY:
Mindfulness is a technique that involves the intentional and non-judgmental regulation of attention to the present moment, with curiosity, openness, and acceptance, as per its definition. Mindfulness-based interventions (MBIs) have been used to manage mood disorders in various clinical and non-clinical settings, including neurological patients and cardiovascular diseases. Studies have consistently demonstrated that MBIs reduce depressive and anxiety symptoms, as well as rumination. MBIs are considered an alternative and effective treatment for reducing psychological stress in the management of different health conditions. Virtual reality (VR) has recently been proposed as an intermediate interface to help patients with emotional dysregulation learn mindfulness practices.

Within this context, new approaches to mental health integrating advanced technologies such as VR can play a critical role. In this interventional study we will seek to demonstrate the effectiveness of a virtual reality-mediated mindfulness-based intervention in a particular group of people who are constantly experiencing psychological distress due to caring for children with autism spectrum disorders (ASD).

DETAILED DESCRIPTION:
In this study participants will be randomly assigned to an experimental or control groups according to the main treatment. Participants in the experimental group will undergo 8 VR sessions by observing a scenario accompanied by a voice audio guide, whereas participants in the control group will complete the 8 VR sessions by observing scenery accompanied only by the sounds of nature. All groups will be treated one time a week for 1h sessions for 8 consecutive weeks.

Participant recruitment: The families of children with ASD will be recruited at the clinical facilities of the Institute for Biomedical Research and Innovation of the National Research Council of Italy (IRIB-CNR) in Messina as part of an ongoing research program.

Allocation of the sample: Eligible participants who will meet the inclusion criteria will receive written information about the procedure and be asked to sign the consent form indicating their willingness to participate in the study. Only qualified individuals who provided informed consent will be randomly assigned to the experimental or control group in a 1:1 manner. Participants will then receive information regarding the allocation result. The randomization will be performed using a computer-generated, site-stratified, randomization schedule. Randomization will be stratified according to age, sex and educational level. For each stratum, random numbers will be assigned to the participants and put into envelopes; it will be determined randomly whether the even or odd number would enter the experimental group. Participants will be assigned to the study according to the numbers they received on opening the envelopes.

Withdrawn criteria: Participants will be considered withdrawn if any of the following occurs: (1) participant chooses to withdraw from the study at any time, (2) intolerable adverse effects, (3) major violation of the study protocol, and (4) other circumstances that would endanger the health of the subject if he/she would to continue his/her participation in the trial.

Immersive virtual environments: Virtual reality experience will be made by using 8 relaxing virtual scenarios (e.g., naturalistic environments) created by BECOME s.r.l. (https://www.discoverbecome.com). The virtual experiences will be offered through the Oculus Quest 2 (marketed since November 2021 as Meta Quest 2)

Sample size: Power size calculation will be performed with GPower 3.1. Considering an anticipated effect size (f) of 1, an alpha set at 0.05, 2 groups, and a 0.95 statistical power, the total sample size required is N = 46.

ELIGIBILITY:
Inclusion Criteria:

* being parent of a child diagnosed with autism
* absence of pharmacotherapy that could interfere with the measured data (psychoactive drugs, anti-hypertensive, anti-depressants)
* no significant visual impairment

Exclusion Criteria:

* history of psychiatric diagnosis
* presence of medical disorders (heart disease or blood pressure, neurological disorders, epilepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Parental Stress Index/Short Form (PSI/SF) | The test needs approximately 10 minutes to complete
  The Parenting Stress Index/Short Form (PSI/SF) is a self-administered questionnaire that aims to identify factors that may negatively impact a child's development
Mindful Attention Awareness Scale (MAAS) | The test needs approximately 10 minutes to complete
  The Mindful Attention Awareness Scale (MAAS) consists of 15 items, each scored on a Likert scale ranging from 1 (almost always) to 6 (almost never). The total score on the MAAS ranges from a minimum of 15 (reflecting a response of 1 on all items) to a maximum of 90 (reflecting a response of 6 on all items). Higher scores on the MAAS indicate greater clinical improvement in a patient's capacity for present moment awareness.
State-Trait Anxiety Inventory (STAI) | The test needs approximately 10 minutes to complete
  The total State-Trait Anxiety Inventory (STAI) score is between 20 and 80 with a predictive threshold value of anxious symptomatology set at 40. The level of severity can also be defined according to a scalar criterion: from 40 to 50 mild form, from 50 to 60 moderate, > of 60 serious.
Beck Depression Inventory (BDI) | The test needs approximately 10 minutes to complete
  The Beck Depression Inventory is a depression rating scale that can be used with individuals 13 years of age and older and assesses symptoms of depression on a scale of 0 to 3 based on 21 specific items.

SECONDARY OUTCOMES:
Heart rate (HR) | The test needs approximately 30 minutes
  The BioHarness 3 uses an electrocardiogram (ECG) sensor to detect the electrical activity of the heart and calculate heart rate in beats per minute (bpm).
Heart rate variability (HRV) | The test needs approximately 30 minutes
  The BioHarness 3 measures the time intervals between successive heart beats and calculates Heart Rate Variability (HRV) in milliseconds (ms).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cerasa, Principal Investigator — antonio.cerasa@irib.cnr.it
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Failla C, Marino F, Bernardelli L, Gaggioli A, Doria G, Chila P, Minutoli R, Mangano R, Torrisi R, Tartarisco G, Bruschetta R, Arcuri F, Cerasa A, Pioggia G. Mediating Mindfulness-Based Interventions with Virtual Reality in Non-Clinical Populations: The State-of-the-Art. Healthcare (Basel). 2022 Jun 29;10(7):1220. doi: 10.3390/healthcare10071220. PMID 35885747
- [Background] Puglisi A, Capri T, Pignolo L, Gismondo S, Chila P, Minutoli R, Marino F, Failla C, Arnao AA, Tartarisco G, Cerasa A, Pioggia G. Social Humanoid Robots for Children with Autism Spectrum Disorders: A Review of Modalities, Indications, and Pitfalls. Children (Basel). 2022 Jun 25;9(7):953. doi: 10.3390/children9070953. PMID 35883937
- [Background] Marino F, Failla C, Carrozza C, Ciminata M, Chila P, Minutoli R, Genovese S, Puglisi A, Arnao AA, Tartarisco G, Corpina F, Gangemi S, Ruta L, Cerasa A, Vagni D, Pioggia G. Mindfulness-Based Interventions for Physical and Psychological Wellbeing in Cardiovascular Diseases: A Systematic Review and Meta-Analysis. Brain Sci. 2021 May 29;11(6):727. doi: 10.3390/brainsci11060727. PMID 34072605